CLINICAL TRIAL: NCT02075645
Title: Can Adherence to PALS Guidelines be Improved by Team Training of Pediatric Resuscitation Members?
Acronym: Teams4Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Elaine Gilfoyle, B.Sc. (Hons.), MD, MMEd, FRCPC, Pediatric Intensivist, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: E-23264
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Crisis Resource Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- team training (Other): Intervention: team training course. A 1-day simulation-based team-training course. There will be 4 simulated resuscitation events. Simulation #1 will be the "pre-course" team performance and simulation #4 will be the "post-course" performance.
  Interventions: Other: Team training course

INTERVENTIONS:
Other: Team training course — A 1-day simulation-based team-training course. There will be 4 simulated resuscitation events. Simulation #1 will be the "pre-course" team performance and simulation #4 will be the "post-course" performance.

SUMMARY:
A multi-centre prospective cohort study, which examines the effect of a team training educational intervention for pediatric resuscitation team members. The study uses simulation-based training as the primary teaching method to evaluate the effect of team training on team performance, as measured by adherence to PALS guidelines. By re-testing participants again after 6-12 months, the study will examine long-term retention of these skills. Hypothesis: adherence to PALS guidelines is improved following team training of pediatric resuscitation team members.

DETAILED DESCRIPTION:
A multi-centre prospective cohort study, which examines the effect of a team training educational intervention for pediatric resuscitation team members. The study uses simulation-based training as the primary teaching method to evaluate the effect of team training on team performance, as measured by adherence to PALS guidelines. By re-testing participants again after 6-12 months, the study will examine long-term retention of these skills.

The investigator anticipates sustained, improved team performance after team training. If this proves to be true, the long-term goal is to disseminate this training widely across Canada, in order to benefit all paediatric resuscitation teams, and ultimately their patients.

ELIGIBILITY:
Inclusion Criteria:

* Code Blue certified RN & RRT
* Pediatric Residents
* Teams must consists of Interprofessional (Resident MD, RN, RRT) resuscitation team members.
* Team composition will reflect actual resuscitation team composition at each site, which will vary slightly from site to site.

Exclusion Criteria:

* Fellows
* Attendings
* Non Code Blue certified staff

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Adherence to PALS guidelines, as measured by the Clinical Performance Tool (CPT) by Donoghue et al | up to 3.5 years

SECONDARY OUTCOMES:
Long-term effect of training on adherence to PALS guidelines (as measured by the CPT) & teamwork performance (as measured by the CTS) at 6-12 months post-training. | up to 3.5 years

OTHER OUTCOMES:
Teamwork performance as measured by the Clinical Teamwork Scale (CTS) by Guise et al | up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Gilfoyle, MD,MMEd, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada